CLINICAL TRIAL: NCT00003540
Title: Phase II Study of Gemcitabine in the Treatment of Patients With Metastatic Breast Cancer Previously Treated With Adriamycin and Taxol
Brief Title: Gemcitabine in Treating Women With Metastatic Breast Cancer Previously Treated With Doxorubicin and Paclitaxel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 98-030; CDR0000066594 (Registry Identifier: PDQ (Physician Data Query)); NCI-G98-1474
Record Dates: First submitted 1999-11-01; First posted 2003-09-25 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine

INTERVENTIONS:
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of gemcitabine in treating women with metastatic breast cancer previously treated with doxorubicin and paclitaxel.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response rate to gemcitabine in women with metastatic breast cancer previously treated with two to four chemotherapy regimens, including doxorubicin and paclitaxel.
* Characterize the nature of toxicity of gemcitabine in this patient population.
* Determine the response duration to gemcitabine in this patient population.

OUTLINE: Patients receive gemcitabine IV over 30 minutes once weekly for 3 consecutive weeks (days 1, 8, and 15) followed by 1 week of rest. Treatment continues every 4 weeks in the absence of disease progression or unacceptable toxic effects.

Patients are followed until death.

PROJECTED ACCRUAL: A total of 14-30 patients will be accrued for this study within 13 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic breast cancer
* Bidimensionally measurable disease

  * No bone scan abnormalities alone
  * Lytic lesions in conjunction with bone scan abnormalities allowed
  * No pure blastic bone metastases
  * No pleural or peritoneal effusions
  * No previously irradiated lesions
* Must have received 2-4 prior chemotherapy regimens, including paclitaxel and doxorubicin, for breast cancer
* Brain metastases allowed if other measurable disease exists

  * No uncontrolled or life threatening brain lesions
* No carcinomatous meningitis
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* AST/ALT no greater than 5 times upper limit of normal

Renal:

* Calcium no greater than 11.0 mg/dL

Other:

* Not pregnant
* Negative pregnancy test
* No history of other malignancy except carcinoma in situ of the cervix or curatively treated nonmelanoma skin cancer
* No other serious medical illnesses, including severe infection and severe malnutrition

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas and mitomycin) and recovered
* No other concurrent chemotherapy

Endocrine therapy:

* Prior hormonal therapies for stage IV disease and/or adjuvant therapy allowed
* At least 3 weeks since prior hormonal therapy

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy to greater than 30% of the marrow bearing bone
* At least 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy to the only measurable lesion

Surgery:

* Recovered from prior surgery
* No concurrent surgery to the only measurable lesion

Other:

* No concurrent nonprotocol treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1998-06; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Violante E. Currie, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States